CLINICAL TRIAL: NCT01786785
Title: Optical Measurement of Cerebral Hemodynamics in Children With Acute Arterial Ischemic Stroke: A Pilot Study
Brief Title: Optical Measurement of Cerebral Hemodynamics in Children With Acute Arterial Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Thrasher Research Fund (Other); National Institutes of Health (NIH) (NIH); Alavi-Dabiri Postdoctoral Fellowship Award (Unknown); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-008442; K12NS049453 (NIH)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Acute Arterial Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stroke Patients: Subjects between 2 and 17 years of age with a confirmed arterial ischemic stroke.
- Controls: Age and Gender Matched Controls

SUMMARY:
Acute ischemic stroke affects roughly 1 in 50,000 children every year and is one of the top ten causes of death in children. Currently, caregivers lay the affected child flat in hopes of increasing blood flow to the brain and reducing the volume of the brain which is damaged. However, there are currently no techniques to measure brain blood flow at the child's bedside and indicate if this treatment is effective. We will probe brain blood volume, oxygen saturation, and flow with red light to determine the efficacy of this intervention.

DETAILED DESCRIPTION:
Arterial ischemic stroke (AIS) affects about 2 children per 100,000 per year and is one of the top 10 causes of mortality in children. After stroke, there is a disturbance in cerebral blood flow (CBF) autoregulation, and changes in head position may change CBF. Currently, practice at the Children's Hospital of Philadelphia (CHOP) is to keep the head of bed (HOB) of a child with AIS flat for 24 hours; however, there is no evidence that this practice is efficacious in children. Furthermore, maintaining a child supine for 24 hours is uncomfortable for the child and is often unenforceable in younger children. This study will use a noninvasive optical technique to measure CBF as HOB position is changed to assess the effectiveness of head of bed position in increasing CBF in children with acute arterial ischemic stroke.

The primary objectives are to determine the difference in CBF at HOB flat (0 degrees) and HOB at +30 degrees in healthy children and in children with AIS. The secondary objectives are to examine CBF in healthy children and in children with AIS at other HOB angles (0, +15, and +30 degrees) compared to the CBF at HOB 0 degrees and to determine if the position that maximizes CBF varies over time from stroke onset.

ELIGIBILITY:
Inclusion Criteria Healthy Control Subjects

1. Subjects age 2-18 years inclusive
2. No history of congenital or acquired brain injury
3. No history of developmental delay, mental retardation, genetic or metabolic syndrome affecting the brain

Inclusion Criteria AIS Subjects

1. Subjects age 2-18 years inclusive
2. 72 hours or less from stroke onset
3. MRI or CT confirmation of AIS

Exclusion Criteria for All Subjects

1. Skull defect preventing application of probes
2. Moyamoya disease
3. Sickle cell anemia

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children (2-18 y.o.) presenting at the Children's Hospital of Philadelphia with a confirmed arterial ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-02; Primary Completion 2016-10-22 (Actual); Study Completion 2016-10-22 (Actual)

PRIMARY OUTCOMES:
Reduction in microvascular blood flow in supine position | 72 hours post stroke
  Microvascular blood flow will be measured at 24, 48, and 72 hours post stroke, with the head of bed at 30, 15, and 0 deg (supine). Current clinical practice is to lower the head of bed to the supine position to increase blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Licht, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States